CLINICAL TRIAL: NCT02611934
Title: Mild Therapeutic Hypothermia for Patients With Acute Coronary Syndrome and Cardiac Arrest Treated With Percutaneous Coronary Intervention
Brief Title: Mild Therapeutic Hypothermia for Patients With Acute Coronary Syndrome and Cardiac Arrest Treated With PCI
Acronym: UNICORN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to insufficient enrollment
Sponsor: Jacek Kubica (Other)
Responsible Party: Sponsor-Investigator, Jacek Kubica, Head of Cardiology, Principal investigator, Collegium Medicum w Bydgoszczy
Organization: Collegium Medicum w Bydgoszczy (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUMK202C
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Arrest; Acute Coronary Syndrome
MeSH Terms: conditions — Heart Arrest; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild Therapeutic Hypothermia (Experimental): OHCA survivors with diagnosed or suspected ACS
  Interventions: Procedure: Mild Therapeutic Hypothermia (MHT)
- no-Mild Therapeutic Hypothermia (No Intervention): OHCA survivors with diagnosed or suspected ACS

INTERVENTIONS:
Procedure: Mild Therapeutic Hypothermia (MHT) — The induction with ice packs and infusion of 0.9% sodium chloride (NaCl) at the temperature of 4˚C. MHT will be maintained with a MTH-dedicated catheter introduced into the inferior vena cava through the femoral vein during PCI. MTH will be maintained for at least 12 hours at target temperature of 33˚C. The rewarming phase will be conducted in an actively controlled manner (0.3˚C per hour). The patient's core temperature will be independently measured in the urinary bladder as well as in the lower one third of the oesophagus using a dedicated catheter and tube. All patients treated with MTH will be mechanically ventilated with a concomitant continuous intravenous infusion of propofol and fentanyl for sedation and analgesia.
  Arms: Mild Therapeutic Hypothermia

SUMMARY:
Mild Therapeutic Hypothermia for Patients with Acute Coronary Syndrome and Cardiac Arrest Treated with Percutaneous Coronary Intervention (UNICORN) study is designed to determine whether mild therapeutic hypothermia (MTH) applied in patients with acute coronary syndromes (ACS) and cardiac arrest treated with percutaneous coronary intervention (PCI) is associated with better clinical outcomes as compared with therapy without MTH.

DETAILED DESCRIPTION:
The UNICORN study is a multi-center, international, observational, phase IV clinical trial which is aimed to investigate whether MTH applied in patients with ACS and cardiac arrest treated with PCI is associated with better clinical outcomes as compared with therapy without MTH. This trial will provide important information regarding the impact of MTH in unconscious with a score of ≤8 on the Glasgow Coma Scale on admission to the hospital after out-of-hospital cardiac arrest (OHCA) with diagnosed or presumed ACS and shockable initial rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Survivor of OHCA
* Sustained return of spontaneous circulation (ROSC) for more than 20 minutes after resuscitation
* Unconsciousness with a score of ≤8 on the Glasgow Coma Scale after ROSC
* Shockable initial rhythm
* Diagnosis or suspicion of ACS

Exclusion Criteria:

* Unwitnessed OHCA
* Obvious or suspected pregnancy
* Known serious infection/sepsis before OHCA
* Known bleeding diathesis
* Confirmed or suspected internal bleeding
* Confirmed or suspected acute stroke
* Confirmed or suspected cerebral injury
* Known serious neurological dysfunction (CPC≤4) before OHCA
* Known serious disease making 180 days of survival unlikely
* Hemodynamic instability with systolic blood pressure <65 mmHg despite treatment
* Time delay from ROSC to MTH induction > 240 min.
* Asystole or pulseless electrical activity (PEA) as the initial rhythm
* Initial body temperature <30°C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 180 days

SECONDARY OUTCOMES:
Neurological outcome according to Cerebral Performance Category (CPC) | at discharge (up to 180 days)
Early stent thrombosis | 30 days
  Definite or confirmed stent thrombosis - symptoms suggestive of an acute coronary syndrome and angiographic or pathologic confirmation of stent thrombosis within 30 days post stent implantation
Bleedings according to the Bleeding Academic Research Consortium (BARC) criteria | 180 days
  bleeding events evaluated based on the BARC definitions
Infectious complications | 180 days
Rhythm and conductions disorders | 180 days
  Rhythm and conductions disorders assessed based on ECG telemetry, 12-lead ECG and ECG holter monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, MD, PhD, Principal Investigator — Collegium Medicum, Nicolaus Copernicus University
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

REFERENCES:
- [Derived] Uminska JM, Ratajczak J, Buszko K, Sobczak P, Sroka W, Marszall MP, Adamski P, Steblovnik K, Noc M, Kubica J. Impact of mild therapeutic hypothermia on bioavailability of ticagrelor in patients with acute myocardial infarction after out-of-hospital cardiac arrest. Cardiol J. 2020;27(6):780-788. doi: 10.5603/CJ.a2019.0024. Epub 2019 Feb 25. PMID 30799546
- [Derived] Uminska JM, Buszko K, Ratajczak J, Lach P, Pstragowski K, Dabrowska A, Adamski P, Skonieczny G, Manitius J, Kubica J. Comparison of temperature measurements in esophagus and urinary bladder in comatose patients after cardiac arrest undergoing mild therapeutic hypothermia. Cardiol J. 2020;27(6):735-741. doi: 10.5603/CJ.a2018.0115. Epub 2018 Sep 24. PMID 30246234
- See also: Study results — https://journals.viamedica.pl/cardiology_journal/article/view/CJ.a2019.0023/47613